CLINICAL TRIAL: NCT00791271
Title: A Parallel Phase I/II Study of Low Dose Decitabine (5-Aza-Deoxycytidine) With Peginterferon Alfa-2b in Advanced Melanoma
Brief Title: Parallel Phase I/II Trial of Decitabine and Peg-Interferon in Melanoma: Phase I Portion
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Schering-Plough (Industry); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0450; NCI-2010-01030 (Registry Identifier: NCI CTRP); NCT02605473 (obsolete NCT alias)
Record Dates: First submitted 2008-11-12; First posted 2008-11-14 (Estimated); Last update posted 2018-11-09 (Actual); Status verified 2018-11

CONDITIONS: Melanoma
Keywords: Melanoma; Malignant melanoma; Unresectable; Decitabine; PEG Interferon Alpha-2b; PEG Intron; 5-Aza-Deoxycytidine; Dacogen
MeSH Terms: conditions — Melanoma | interventions — Decitabine; peginterferon alfa-2b

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Decitabine + Peginterferon Alfa-2b (Experimental): Decitabine starting dose of 10mg/m^2 given daily via intravenous infusion on days 1-5 of 28 day cycle. Peginterferon Alfa-2b starting dose of 3 µg/kg injection under the skin once a week on days 1, 8, 15, and 21 of 28 day cycle.
  Interventions: Drug: Decitabine; Drug: Pegylated Interferon Alpha-2b

INTERVENTIONS:
Drug: Decitabine — Starting dose of 10mg/m^2 given daily via intravenous infusion on days 1-5 of 28 day cycle.
  Other Names: 5-Aza-Deoxycytidine; Dacogen
Drug: Pegylated Interferon Alpha-2b — Starting dose of 3 µg/kg injection under the skin once a week on days 1, 8, 15, and 21 of 28 day cycle.
  Other Names: PEG Interferon Alpha-2b; PEG Intron

SUMMARY:
The goal of the first phase of this clinical research study is to find the highest tolerable dose of decitabine and peginterferon alfa-2b that can be given in combination to patients with melanoma. The safety of this drug combination will also be studied.

The goals of the second phase are to learn if decitabine and peginterferon alfa-2b combined can help to control melanoma, and to find out which doses are more effective and/or better tolerated.

DETAILED DESCRIPTION:
The Study Drugs:

Decitabine is designed to damage the DNA of cells, which may cause cancer cells to die.

Peginterferon alfa-2b is designed to strengthen the immune system, which may decrease tumor growth.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you joined this study. Up to 6 groups of 3-6 participants will be enrolled in the Phase I portion of the study, and up to 44 participants will be enrolled in Phase II.

If you are enrolled in the Phase I portion, the dose of decitabine and peginterferon alfa-2b you receive will depend on when you joined this study. The first group of participants will receive the lowest dose level of the study drug combination. Each new group will receive a higher dose level than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of the study drug combination is found.

If you are enrolled in the Phase II portion, the dose of decitabine and peginterferon alfa-2b you receive will depend on when you joined this study, as well as the research data from the Phase I portion. You will be randomly assigned (as in the roll of dice) to receive one of the dose levels (which may be from 1 to 6 dose levels, depending on the available data from the Phase I portion) that have been found in the Phase I portion to have the least side effects and to be possibly the most effective. This means you will have an equal chance of being assigned to any of the dose levels that are being used at that time. As the study goes on, if the research data suggests that one dose level may be better tolerated than the others, new participants enrolling into the Phase II portion would be more likely to be assigned to that possibly better dose level.

No matter which phase you are enrolled in, your dose of the study drugs may be lowered if you do not tolerate the study drug combination well.

Study Drug Administration:

A "cycle" on this study is 28 days. Decitabine will be given by vein, over 1 hour, on Days 1-5 of each cycle. Peginterferon alfa-2b will be given by injection under the skin, once a week (on Days 1, 8, 15, and 21). You will be giving peginterferon alfa-2b to yourself under nursing supervision on the days you are receiving decitabine.

On Day 6 of each cycle, you will either receive Neulasta (pegfilgrastim) or Neupogen (filgrastim). Pegfilgrastim or filgrastim will be injected under your skin. If you receive pegfilgrastim, it will be injected only on Day 6 of each cycle. If you receive filgrastim, it will be injected 1 time a day for as many days as the doctor decides is needed to raise your white blood cell count.

Study Visits:

On Day 1 of each cycle, the following procedures will be performed:

* You will have a physical exam, including measurement of your vital signs and weight.
* You will be asked about any medications or treatments you may be currently receiving and any side effects you may have experienced.
* You will have a performance status evaluation.
* Blood (about 1 teaspoon) will be drawn for routine tests.

These same tests listed above will be repeated at additional visits with the research nurse during Week 3 of Cycles 1 and 2. If you do not experience severe side effects during Cycles 1 and 2, these extra Week 3 visits with the research nurse will no longer be necessary in later cycles. They may, however, be started again if needed.

At the end of of Cycle 3, and every odd cycle after that (Cycles 5, 7, 9, and so on), you will have a scan performed (such as CT or MRI) to check the status of the disease.

Length of Study Participation:

You may remain on study for as long as you are benefitting. If the disease gets worse or intolerable side effects occur, you will be taken off study early.

End-of-Study Visit:

Once you go off study for any reason, you will have an end-of-study visit with the same procedures performed as the Day 1 study visits. You may also have a scan performed (such as CT or MRI) to check the status of the disease if you have not had one performed in the last 4 weeks.

Long-Term Follow-Up:

Every 3 months for about 2 years, researchers will call you to see how you are doing.

This is an investigational study. Decitabine is FDA approved and commercially available for the treatment of myelodysplastic syndrome (MDS). Peginterferon alfa-2b is FDA approved and commercially available for the treatment of hepatitis C. Their use together in this study in the treatment of melanoma is considered experimental. At this time, the combination is being used in research only.

Up to 80 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have pathologically confirmed malignant melanoma that is unresectable stage III or stage IV.
2. Patients must have measurable disease as defined by RECIST criteria.
3. No more than two prior chemotherapy for unresectable stage III or IV melanoma.
4. Patients must be >/= 28 days beyond the last administration of anticancer therapy, and must have recovered from the toxicities of prior therapy. If the patient was recently treated with a nitrosurea, they must be >/= 42 days beyond the last administration.
5. Patients must have no other active malignancies. Patients with prior history of any in situ cancer, lobular carcinoma of the breast in situ, cervical cancer in situ, atypical melanocytic hyperplasia or Clark I melanoma in situ or basal or squamous cell skin cancer are eligible. Patients with other malignancies are eligible, if their disease has been inactive for 2 years prior to the time of study entry.
6. Patients must be >/= 18 years of age.
7. Patients must give written informed consent prior to initiation of therapy in keeping with the policies of the institution. Patients with a history of major psychiatric illness must be judged able to fully understand the investigational nature of this study and the risks associated with the therapy.
8. Women of childbearing potential (WOCBP) must not be pregnant (negative urine human chorionic gonadotropin (HCG) within 2 weeks of treatment) or lactating. A WOCBP is defined as a woman who has not undergone a hysterectomy or who has had menses at any time in the preceding 24 consecutive months.
9. Women of childbearing potential and sexually active males must be counseled to use an accepted and effective method of contraception (including abstinence) while on treatment and for a period of 3 months after completing or discontinuing treatment.
10. Patients must have Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
11. Patients must have adequate organ and marrow function, measured within 14 days of study entry, as defined below: All Patients: - Absolute neutrophil count >/=1,500/uL - Platelets >/=100,000/uL - Creatinine (serum) </= 2.0 mg/dL - Total bilirubin </= 1.5 mg/dL - AST(SGOT)/ALT(SGPT) </= 2.5 X Institutional Upper Limit of Normal (IULN)
12. Patients with any number of prior targeted or cytokine therapies, but no more than two chemotherapy containing regimens.

Exclusion Criteria:

1. Patients with active autoimmune disorders or who are receiving immunosuppressive therapy (including steroids or methotrexate) for any indication are excluded. An exception may be made, by the PI, to include patients with adrenal insufficiency requiring physiologic steroid hormone replacement only.
2. Patients who have previously received adjuvant high dose interferon.
3. Patients may not receive any other investigational agents within four weeks of study entry. Patients may not receive any other investigational agents while on study.
4. Patients who have had major surgery within 2 weeks prior to entering the study, or have otherwise not adequately recovered from prior surgery.
5. Patients who have had palliative radiation therapy within 2 weeks prior to entering the study.
6. Patients with brain metastases.
7. Patients with a history of active ischemic heart disease or cerebro-vascular disease, congestive heart failure (NYHA class >2) or anginal syndrome requiring ongoing medical treatment.
8. Patients with myocardial ischemia (MI), stroke, or transient ischemic attack (TIA) within the last 6 months.
9. Patients with a diagnosis or evidence of organic brain syndrome or significant impairment of basal cognitive function or any psychiatric disorder that might preclude participation in the protocol.
10. Patients with a history of central nervous system (CNS) demyelinating, inflammatory disease or hereditary or acquired peripheral neuropathy.
11. Patients with known history of HIV and hepatitis infection or any other significant medical or surgical condition or psychiatric disorder that may interfere with the completion of this trial or with the evaluation of safety and efficacy of the study combination.
12. Patients with thyroid dysfunction not responsive to therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09-02 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Phase I: Dose-limiting toxicity (DLT) | 4 weeks
  Dose limiting toxicity defined as any treatment related toxicity that meets one or more of the following criteria:
  Any grade 3 or 4 non-hematologic toxicity regardless of duration, except:
  1. Grade 3 nausea or vomiting occurring without maximal antiemetic therapy.
  2. Grade 3 diarrhea that occurs following without adequate loperamide therapy.
     * Grade 4 thrombocytopenia.
     * Grade 4 neutropenia lasting > 2 weeks or associated with infection.
     * Any toxicity that results in a treatment delay of > 4weeks.

SECONDARY OUTCOMES:
Phase II: Patient Response | 12 weeks
  Success defined as either a complete response (CR), a partial response (PR), or stable disease (SD). Target combined endpoint of CR+PR+SD in this trial is 30%. Evaluation of response follows the Response Evaluation Criteria in Solid Tumors (RECIST) Guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Jen Hwu, MD, PhD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org